CLINICAL TRIAL: NCT00149227
Title: Add-on Effects of Valsartan on Morbi- Mortality in High Risk Hypertension
Brief Title: Add-on Effects of Valsartan on Morbi- Mortality (KYOTO HEART Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyoto Prefectural University of Medicine (Other)
Responsible Party: Principal Investigator, Hiroaki Matsubara, MD., PhD, Add-on Effects of Valsartan on Morbi- Mortality in High Risk Hypertension, Kyoto Prefectural University of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KHS2004
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Hypertension; Ischemic Heart Disease; Congestive Heart Failure; Stroke
Keywords: High risk hypertension; Ischemic heart disease; Angiotensin receptor blockers; Cardiovascular mortality- morbidity; KYOTO HEART Study
MeSH Terms: conditions — Hypertension; Myocardial Ischemia; Heart Failure; Stroke | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-ARB (Active Comparator): 'Non-ARB' was defined as Conventional anti-hypertensive treatment except for ARB and ACEIs
  Interventions: Drug: Non-ARB
- Valsartan (Experimental): Valsartan add-on treatment
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Valsartan — Valsartan add-on arm: valsartan 40-160 mg per day, and an additional antihypertensive drugs other than ARB and ACEI are administered if necessary.
  Other Names: Diovan
  Arms: Valsartan
Drug: Non-ARB — 'Non-ARB' was defined conventional anti-hypertensive treatment except for ACEIs and ARBs
  Other Names: Conventional anti-hypertensive treatment
  Arms: Non-ARB

SUMMARY:
The KYOTO HEART Study is to assess the add-on effect of valsartan, an Angiotensin-Receptor Blocker, on top of the conventional treatment in high risk patients in Japan with hypertension in terms of the morbidity and mortality.

DETAILED DESCRIPTION:
Although many reports show that ACE inhibitors and angiotensin II receptor blockers (ARB) are superior for prevention of cardiovascular events, previous data are not enough for the patients who have more than one risk factor and for anti-atherosclerotic effects of ARB. In Japan, there were only a few large-scale trials for cardiovascular disease prevention, and it has not been clarified whether the evidence in Western countries could be unqualifiedly applied to Japanese patients as a long-range strategy. The KYOTO HEART Study is to assess the add-on effect of valsartan, an Angiotensin-Receptor Blocker, on top of the conventional treatment in high risk patients with hypertension in terms of the morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension
* Clinical diagnosis of one or more risk factors, such as diabetes, smoking habit, lipid metabolism abnormality, history of ischemic heart disease (IHD) or cerebrovascular disease, obesity (BMI>25), chronic heart failure (NYHA II-III), and electrocardiogram (ECG) abnormality (LVH)

Exclusion Criteria:

* Patients who have already been administered ARB
* Patients with IHD within 6 months after percutaneous coronary intervention(PCI), and who are stable but are going to implement PCI or coronary artery bypass grafting(CABG)
* Severe/malignant/secondary hypertensive patients
* Pregnant women and women of childbearing potential
* History of heart failure, unstable angina, myocardial infarction, PTCA, or CABG within the preceding 6 months
* Arrhythmia needed to be treated or accompanied with symptoms, second or third degree AV block
* Severe renal impairment (Serum creatinine >3.0 mg/dl)
* Severe hepatic impairment (Hepatic failure, Cirrhosis, etc.)

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3031 (Actual)
Dates: Start 2004-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Matsubara, MD,PhD, Study Chair — Kyoto Prefectural University of Medicine
Locations (1):
- Kyoto Prefectural University of Medicine, Kyoto, Kyoto, Japan

REFERENCES:
- [Background] Sawada T, Takahashi T, Yamada H, Dahlof B, Matsubara H; KYOTO HEART Study Group. Rationale and design of the KYOTO HEART study: effects of valsartan on morbidity and mortality in uncontrolled hypertensive patients with high risk of cardiovascular events. J Hum Hypertens. 2009 Mar;23(3):188-95. doi: 10.1038/jhh.2008.116. Epub 2008 Sep 18. PMID 18800142
- [Result] Sawada T, Yamada H, Dahlof B, Matsubara H; KYOTO HEART Study Group. Effects of valsartan on morbidity and mortality in uncontrolled hypertensive patients with high cardiovascular risks: KYOTO HEART Study. Eur Heart J. 2009 Oct;30(20):2461-9. doi: 10.1093/eurheartj/ehp363. Epub 2009 Aug 31. PMID 19723695 (Retraction: PMID 23376450 Eur Heart J. 2013 Apr;34(14):1023)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited patients between January 2004 and June 2007. Participating centres included 31 associated hospitals led by physicians (cardiology specialists) from Kyoto Prefectural University School of Medicine.
Pre-assignment Details: Among 3042 patients eligible, 4 patients were withdrawn due to refusal of informed consent, 7 were withdrawn due to incompatible object. Finally, 3031 patients were assigned to the treatment groups.
Groups:
- Valsartan: For the valsartan add-on group, valsartan 80 mg once daily in the morning was administered to the patient as an initial dose, the dose was doubled after 4 weeks if the initial dose could not achieve the target blood pressure of less than 140/90 mmHg (in patients with diabetes or renal disease, target blood pressure was set to less than 130/80 mmHg). After 8 weeks, an additional administration of other antihypertensive drugs with ﬂexible dosing regimen other than ARBs and ACE inhibitors was allowed if necessary.
- Non-ARB: For the conventional treatment group, the anti-hypertensive drugs other than ARB and ACE inhibitors were provided for the patients to reach the target blood pressure.
Period: Overall Study
Arm/Group | Valsartan | Non-ARB
Started | 1517 | 1514
Completed | 1517 | 1514
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan | Non-ARB | Total
Number analyzed (Participants) | 1517 | 1514 | 3031
Age Continuous [Mean (Standard Deviation); unit: years] | 65.8 (11.2) | 66.1 (10.9) | 65.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 656 | 647 | 1303
  Male | 861 | 867 | 1728
Region of Enrollment [Number; unit: participants]
  Japan | 1517 | 1514 | 3031

OUTCOME MEASURES:

1. Primary Outcome: New Onset or Recurrence of Stroke
Description: Stroke events included brain hemorrhage, infarction, and TIA. They required hospitalization with neurological symptoms and were diagnosed by CT and/or MRI. The first of any of these events to occur in a specific patient was classified as an event to be counted in the primary endpoint by the Endpoint Committee. We estimated the number of enrolled patients to validate the hypothesis under the assumption that the valsartan add-on group achieves a 20% risk reduction compared with the conventional treatment group and gives 80% statistical power for detecting a clinical signiﬁcance with a two-tailed 5% statistical signiﬁcant level.
Time Frame: five years
Population: Analyses were made by the independent Statistical Analysis Organization based on the intention-to-treat principle.
Measure: Number; unit: event number
Arm/Group | Valsartan | Non-ARB
Number analyzed (Participants) | 1517 | 1514
event number | 25 | 46
Statistical Analysis 1: Comparison: Valsartan vs Non-ARB; We estimated the number of enrolled patients to validate the hypothesis under the assumption that the valsartan add-on group achieves a 20% risk reduction compared with the conventional treatment group and gives 80% statistical power for detecting a clinical signiﬁcance with a two-tailed 5% statistical signiﬁcant level. with a two-tailed 5% statistical signiﬁcant level; Test type: Superiority or Other; p < 0.05, Cox's proportional hazard analysis; Cox Proportional Hazard = 0.8, 95% CI 2-sided [-0.975 to 0.975], Standard Deviation 2

2. Primary Outcome: New Onset or Recurrence of Transient Ischemic Attack
Description: Transient ischemic attack (TIA) was defined as hospitalization with sudden onset of neurological deficit persisting for less than 24 hrs, and without abnormal findings using by CT and/or MRI. The first of any of these events to occur in a specific patient was classified as an event to be counted in the primary endpoint by the Endpoint Committee. We estimated the number of enrolled patients to validate the hypothesis under the assumption that the valsartan add-on group achieves a 20% risk reduction compared with the conventional treatment group and gives 80% statistical power for detecting a clinical signiﬁcance with a two-tailed 5% statistical signiﬁcant level.
Time Frame: five years
Measure: Number; unit: event number
Arm/Group | Valsartan | Non-ARB
Number analyzed (Participants) | 1517 | 1514
event number | 6 | 4

3. Primary Outcome: New Onset or Recurrence of Acute Myocardial Infarction
Description: Acute myocardial infarction was diagnosed with hospitalization, ECG- change, and biomarkers for myocardial infarction. The first of any of these events to occur in a specific patient was classified as an event to be counted in the primary endpoint by the Endpoint Committee. We estimated the number of enrolled patients to validate the hypothesis under the assumption that the valsartan add-on group achieves a 20% risk reduction compared with the conventional treatment group and gives 80% statistical power for detecting a clinical signiﬁcance with a two-tailed 5% statistical signiﬁcant level.
Time Frame: five years
Measure: Number; unit: event number
Arm/Group | Valsartan | Non-ARB
Number analyzed (Participants) | 1517 | 1514
event number | 7 | 11

4. Primary Outcome: Hospitalization Due to the New Onset, Recurrence or Worsening of Heart Failure and Additional Concomitant Use of Other Anti-heart Failure Agents or Increase of Dosage
Description: Heart failure event was defined as requiring hospitalization and clinical symptoms together with left ventricular dysfunction by echocardiography according to the guidelines of the AHA/ACC. The first of any of these events to occur in a specific patient was classified as an event to be counted in the primary endpoint by the Endpoint Committee. We estimated the number of enrolled patients to validate the hypothesis under the assumption that the valsartan add-on group achieves a 20% risk reduction compared with the conventional treatment group and gives 80% statistical power for detecting a clinical signiﬁcance with a two-tailed 5% statistical signiﬁcant level.
Time Frame: five years
Measure: Number; unit: event number
Arm/Group | Valsartan | Non-ARB
Number analyzed (Participants) | 1517 | 1514
event number | 12 | 26

5. Primary Outcome: Hospitalization Due to the New Onset, Occurrence or Worsening of Angina Pectoris and Additional Concomitant Use of Other Anti-anginal Agents or Increase of Dosage
Description: Angina pectoris event required hospitalization and was diagnosed by both ECG changes corresponding with chest symptoms and coronary angiography showing 75% stenosis according to AHA/ACC guidelines. The first of any of these events to occur in a specific patient was classified as an event to be counted in the primary endpoint by the Endpoint Committee. We estimated the number of enrolled patients to validate the hypothesis under the assumption that the valsartan add-on group achieves a 20% risk reduction compared with the conventional treatment group and gives 80% statistical power for detecting a clinical signiﬁcance with a two-tailed 5% statistical signiﬁcant level.
Time Frame: five years
Measure: Number; unit: event number
Arm/Group | Valsartan | Non-ARB
Number analyzed (Participants) | 1517 | 1514
event number | 22 | 44

6. Primary Outcome: Operation of PCI or Bypass Operation
Time Frame: five years
Reporting Status: Not Posted
Measure: Number; unit: event number

7. Primary Outcome: New Onset of Acute Dissecting Aneurysm of the Aorta
Description: Dissecting aneurysm of the aorta required hospitalization and was diagnosed by imaging technique, CT and/or MRI. The first of any of these events to occur in a specific patient was classified as an event to be counted in the primary endpoint by the Endpoint Committee. We estimated the number of enrolled patients to validate the hypothesis under the assumption that the valsartan add-on group achieves a 20% risk reduction compared with the conventional treatment group and gives 80% statistical power for detecting a clinical signiﬁcance with a two-tailed 5% statistical signiﬁcant level.
Time Frame: five years
Measure: Number; unit: event number
Arm/Group | Valsartan | Non-ARB
Number analyzed (Participants) | 1517 | 1514
event number | 3 | 5

8. Primary Outcome: New Onset, Recurrence or Worsening of Arteriosclerosis Obliterans
Description: Arteriosclerosis obliterans (ASO) event was diagnosed with symptoms and CT / MRI imaging. The first of any of these events to occur in a specific patient was classified as an event to be counted in the primary endpoint by the Endpoint Committee. We estimated the number of enrolled patients to validate the hypothesis under the assumption that the valsartan add-on group achieves a 20% risk reduction compared with the conventional treatment group and gives 80% statistical power for detecting a clinical signiﬁcance with a two-tailed 5% statistical signiﬁcant level.
Time Frame: five years
Measure: Number; unit: event number
Arm/Group | Valsartan | Non-ARB
Number analyzed (Participants) | 1517 | 1514
event number | 11 | 12

9. Primary Outcome: Transition to Dialysis, Doubling of Plasma Cr Levels
Description: The first of any events, "transition to dialysis" or "doubling of plasma Cr levels compared to the entry", occurring in a specific patient was classified as an event to be counted in the primary endpoint by the Endpoint Committee. We estimated the number of enrolled patients to validate the hypothesis under the assumption that the valsartan add-on group achieves a 20% risk reduction compared with the conventional treatment group and gives 80% statistical power for detecting a clinical signiﬁcance with a two-tailed 5% statistical signiﬁcant level.
Time Frame: five years
Measure: Number; unit: event number
Arm/Group | Valsartan | Non-ARB
Number analyzed (Participants) | 1517 | 1514
event number | 6 | 14

10. Secondary Outcome: All Cause Mortality
Time Frame: five years
Measure: Number; unit: patients
Arm/Group | Valsartan | Non-ARB
Number analyzed (Participants) | 1517 | 1514
patients | 22 | 32

11. Secondary Outcome: Worsening of Cardiac Function
Time Frame: five years
Reporting Status: Not Posted
Measure: Number; unit: event number

12. Secondary Outcome: New Onset or Worsening of Arrhythmias
Time Frame: five years
Reporting Status: Not Posted
Measure: Number; unit: event number

13. Secondary Outcome: New Onset or Worsening of Diabetes Mellitus or IGT
Description: Diabetes mellitus was defined as fasting plasma glucose >=126 mg/dl, causal blood glucose >= 200 mg /dl, HbA1C >= 6.5%, and/or plasma glucose 2hr after 75g glucose load >= 200 mg/dl. The first of these events, "new onset diabetes" or "worsening diabetes following IGT", occurring in a specific patient was classified as an event to be counted in the secondary endpoint by the Endpoint Committee. We estimated the number of enrolled patients to validate the hypothesis under the assumption that the valsartan add-on group achieves a 20% risk reduction compared with the conventional treatment group and gives 80% statistical power for detecting a clinical signiﬁcance with a two-tailed 5% statistical signiﬁcant level.
Time Frame: five years
Measure: Number; unit: event number
Arm/Group | Valsartan | Non-ARB
Number analyzed (Participants) | 1517 | 1514
event number | 58 | 86

14. Secondary Outcome: Uncontrolled Blood Pressure, Etc.
Time Frame: five years
Reporting Status: Not Posted
Measure: Number; unit: patients

ADVERSE EVENTS:
Arm/Group | Valsartan | Non-ARB
Serious Adverse Events (participants affected / at risk) | 0/1517 | 0/1514
Other Adverse Events (participants affected / at risk) | 0/1517 | 0/1514

LIMITATIONS AND CAVEATS:
The study was performed using PROBE design, which does not exclude possible bias for softer endpoints such as angina and TIA. However, all softer endpoints were diagnosed by CAG and CT/MRI. We believe that under reporting would be unlikely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No